CLINICAL TRIAL: NCT01238393
Title: A Prospective Pilot Study of Lucentis for Epiretinal Membranes: the LERM Study
Brief Title: Treatment of Epiretinal Membranes With Ranibizumab
Acronym: LERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTH-092-10
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental): ('intravitreal ranibizumab' )
  Interventions: Drug: intravitreal ranibizumab

INTERVENTIONS:
Drug: intravitreal ranibizumab — monthly injections x3 +/- 2nd series of 3
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to determine whether intraocular injection of ranibizumab decreases the retinal thickness in patients with epiretinal membranes and reduces associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic idiopathic epiretinal membrane

Exclusion Criteria:

* vision worse than 6/18 and fit for surgery
* prior vitreoretinal surgery or injection
* diabetes
* any past or current form of retinal vein occlusion or neovascularization
* age-related macular degeneration
* other condition causing significant limitation of visual potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Evidence of improvement measured by optical coherence tomography | 3 and 6 months

SECONDARY OUTCOMES:
Distance visual acuity (ETDRS) | 3 and 6 months
Near visual acuity (Snellen) | 3 and 6 months
Subjective change in symptoms | 3 and 6 months
Amsler grid improvement | 3 and 6 months
Quality of life improvement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gale, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Hotel Dieu Hospital, Kingston, Ontario, Canada